CLINICAL TRIAL: NCT01547481
Title: Statistical Mapping of the Brain in Progressive Supranuclear Palsy, Essential Tremor, Parkinson Disease, Parkinsonism, and REM Behavior Disorder
Brief Title: MRI Study of Brain Activity in Healthy Adults and Individuals With Parkinsonism and Rapid Eye Movement Disorder.
Status: Completed | Type: Observational
Sponsor: University of Alabama at Birmingham (Other)
Responsible Party: Principal Investigator, Dr. Frank Michael Skidmore, Assistant Professor, University of Alabama at Birmingham
Other Study IDs: fMRI - Skidmore
Record Dates: First submitted 2012-02-28; First posted 2012-03-07 (Estimated); Last update posted 2018-05-17 (Actual); Status verified 2018-05

CONDITIONS: Movement Disorders (Incl Parkinsonism); Tremor Familial Essential, 1; REM Sleep Behavior Disorder
MeSH Terms: conditions — Movement Disorders; Tremor hereditary essential, 1; REM Sleep Behavior Disorder

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (6):
- Parkinson's Disease Cohort: Individuals Diagnosed with Parkinson's Disease
- Essential Tremor cohort: Individuals Diagnosed with Essential Tremor
- Rapid Eye Movement Disorder Cohort: Individuals Diagnosed with Rapid-Eye Movement Behavior Disorder (RBD). Eligible individuals will have been diagnosed with RBD based on a sleep study prior to entering the study. This study does not pay for or support a sleep study.
- Healthy Control group: Individuals are healthy, without a known neurologic disease.
- Progressive Supranuclear Palsy Cohort: Individuals diagnosed with Progressive Supranuclear Palsy (PSP).
- Parkinsonism - Undifferentiated: Individuals with any form of Parkinsonism, not meeting any of the above cohorts.

SUMMARY:
This proposal is focused on developing a reliable, valid, and reproducible imaging techniques and statistical methodology for segregation of various forms of Parkinsonism from healthy adults without Parkinsonism.

DETAILED DESCRIPTION:
This proposal is focused on developing a reliable, valid, and reproducible imaging techniques and statistical methodology for segregation of various forms of Parkinsonism from healthy adults without Parkinsonism. We focus on early diagnosis of Parkinsonism, other tremor disorders, and determine how imaging might be used to improve diagnosis. The purpose of this protocol is to gather a multi-modal dataset to explore and validate the investigator's previous research findings in prior studies.

ELIGIBILITY:
Inclusion Criteria:

* Healthy Control • Age 35-85

Parkinson Disease (PD) Age 35-85

Diagnosis of clinically definite PD made by a movement disorders specialist, with evidence of the following features:

* Presence of bradykinesia and 1 or both of the following:

  1. Rest tremor
  2. Rigidity
* Asymmetric Onset
* Progressive motor symptoms
* Levodopa responsive
* Duration at least 1 but not more than 10 years
* Hoehn and Yahr Stage 1-2

Progressive Supranuclear Palsy (PSP) Age 40-85

Diagnosis of clinically definite PSP, with the following features:

* Gradually progressive disorder.
* Onset after age 39
* Supranuclear palsy* and postural instability with falls in the first year of disease onset*.
* No evidence of other disease.

Parkinsonism of Other or Undetermined Cause (POC) Age 35-85

Diagnosis of parkinsonism of undetermined other other cause by a movement disorders specialist, with the following features:

* Signs and symptoms of Parkinsonism including

  1. Bradykinesia
  2. Mixed or resting tremor
  3. Rigidity
  4. Characteristic deficits of gait and balance associated with Parkinsonism

     Essential Tremor (ET) Age 35-85

     Diagnosis of essential tremor, with the following features:
* A 2+ postural tremor of at least 1 arm (a head tremor may also be present, but is not sufficient for diagnosis)
* On examination, there must be

  1. a 2+ kinetic tremor during at least 4 tasks, or;
  2. a 2+ kinetic tremor on 1 task and a 3+ kinetic tremor on a second task; tasks include pouring water, using a spoon to drink water, drinking water, finger-to-nose, and drawing a spiral
* If on examination, the tremor is present in the dominant hand, then by report, it must interfere with at least 1 activity of daily living.

REM Behavior Disorder (RBD) Age 25 - 85

Documented diagnosis of REM sleep behavior disorder (RBD) by a sleep medicine specialist, with the following clinical features:

* Presence of REM sleep without atonia on polysomnography
* At least one of the following conditions:

  1. Sleep-related, behaviors by history (eg, dream enactment behavior)
  2. Abnormal REM sleep behavior documented during PSG monitoring

Exclusion Criteria:

Healthy Control

* Pregnancy
* First-degree blood relative affected by PD
* Neurodegenerative disease
* History of repeated head injury, encephalitis, brain surgery, stroke, dementia, neuroleptic exposure, or serious medical illness that may interfere with participation.

Parkinson Disease (PD)

* Any exclusion criteria that would exclude a healthy control patient
* Atypical features indicative of a Parkinson-Plus disorder

Progressive Supranuclear Palsy (PSP)

* Any exclusion criteria that would exclude a healthy control patient
* Any finding atypical for PSP
* Neuroradiologic evidence of relevant structural abnormality unrelated to appropriate changes known to be associated with PSP

Parkinsonism of Other or Undetermined Cause (POC)

* Any exclusion criteria that would exclude a healthy control patient
* Signs and symptoms suggestive of clear diagnosis of idiopathic Parkinson disease, Progressive Supranuclear Palsy, or Essential Tremor

Essential Tremor (ET)

* Any exclusion criteria that would exclude a healthy control patient
* No other potential etiologic factors for the tremor
* Any first-degree blood relative affected by PD
* History of neurodegenerative disease

REM Behavior Disorder (RBD)

* Any exclusion criteria that would exclude a healthy control patient
* Sleep disorder not better explained by another sleep disorder, medical or neurological disorder, mental disorder, medication use, or substance use disorder

Ages: 19 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Subjects with PD, MSA-P, ET, or PSP will be recruited based on clinical criteria from the UAB Comprehensive Parkinson Disease and Movement Disorder Clinic located at The Kirklin Clinic at UAB. This center sees over 3,500 patients annually. Individuals with RBD will be recruited from the UAB University Hospital and UAB Highlands Sleep Disorders Center and will be identified through patient contact with a UAB Department of Neurology physician.
Sampling Method: Non-Probability Sample
Enrollment: 50 (Actual)
Dates: Start 2011-12; Primary Completion 2015-12-31 (Actual); Study Completion 2015-12-31 (Actual)

PRIMARY OUTCOMES:
fMRI compared between cohorts | one time at initial visit
  Studying resting brain activity between healthy adults, participants with Parkinson's and participants with REM Behavior Disorder.

CONTACTS AND LOCATIONS:
Overall Officials: Frank Skidmore, MD, Principal Investigator — University of Alabama at Birmingham
Locations (1):
- University of Alabama at Birmingham, Birmingham, Alabama, United States

IPD SHARING:
Plan to Share IPD: Yes
Patient data has now been collated as a de-identified dataset, that can be shared if requested.